CLINICAL TRIAL: NCT05698472
Title: A Study on the Status Quo of Physical Exercise for the Elderly in Beijing Community
Brief Title: A Study on the Status Quo of Physical Exercise for the Elderly
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: M2022735
Record Dates: First submitted 2023-01-16; First posted 2023-01-26 (Actual); Last update posted 2023-01-26 (Actual); Status verified 2022-11

CONDITIONS: Physical Exercise; Elderly; Community
MeSH Terms: conditions — Motor Activity | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: questionnaire — Use the "Questionnaire on physical exercise of the elderly in Beijing community" to collect the related information of the elderly.

SUMMARY:
Through interview, taking the elderly community in Beijing as an example, this study will try to further understand the current physical exercise situation of the elderly in the community, and analyze the factors influencing their participation degree. By this way, we will try to provide constructive suggestions for the development and design of universal community physical exercise programs for the elderly.

ELIGIBILITY:
Inclusion Criteria:

1. Regardless of gender, age ≥ 65 years old
2. Lived in Beijing for a long time
3. Normal listening, speaking, and comprehension skills

Exclusion Criteria:

1. Accompanied by significant cognitive dysfunction
2. Diseases that seriously affect their participation in sports, such as fractures, tumors, neurological diseases, etc.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: The elderly who has lived in Beijing for a long period and is older than 65 years old.
Sampling Method: Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2022-11-25 (Actual); Primary Completion 2023-01-02 (Actual); Study Completion 2023-02-25 (Estimated)

PRIMARY OUTCOMES:
questionnaire | 1 day (once)
  Use the "Questionnaire on physical exercise of the elderly in Beijing community" to collect the related information of the elderly.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University Third Hospital, Beijing, Beijing Municipality, China